CLINICAL TRIAL: NCT05547464
Title: A Phase Ib/IIa Two-part, Randomized, Placebo-controlled, Observer-blind, Dose-finding Evaluation Trial to Describe the Safety, Reactogenicity, and Immunogenicity of Two Investigational Vaccines Against Tuberculosis in BCG Vaccinated, HIV-negative Subjects
Brief Title: Safety and Immune Responses After Vaccination With Two Investigational RNA-based Vaccines Against Tuberculosis in BCG Vaccinated Volunteers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BNT164-02; DOH-27-052023-8662 (Registry Identifier: SANCTR); PACTR202505818080160 (Registry Identifier: PACTR)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis
Keywords: Prevention of tuberculosis; RNA Vaccine; Vaccine; TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A: BNT164a1 (Experimental): Escalating dose levels
  Interventions: Biological: BNT164a1
- Part A: BNT164b1 (Experimental): Escalating dose levels
  Interventions: Biological: BNT164b1
- Part B: BNT164a1 Dose level (DL) 1 (Experimental)
  Interventions: Biological: BNT164a1
- Part B: BNT164a1 DL 2 (Experimental)
  Interventions: Biological: BNT164a1
- Part B: BNT164b1 DL 1 (Experimental)
  Interventions: Biological: BNT164b1
- Part B: BNT164b1 DL 2 (Experimental)
  Interventions: Biological: BNT164b1
- Placebo (Placebo Comparator): Isotonic sodium chloride (NaCl) solution (0.9%)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT164a1 — Multi-antigen ribonucleic acid (RNA) vaccine for active immunization against tuberculosis administered as intramuscular injection
  Arms: Part A: BNT164a1; Part B: BNT164a1 DL 2; Part B: BNT164a1 Dose level (DL) 1
Biological: BNT164b1 — Multi-antigen RNA vaccine for active immunization against tuberculosis administered as intramuscular injection
  Arms: Part A: BNT164b1; Part B: BNT164b1 DL 1; Part B: BNT164b1 DL 2
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a two-part randomized, placebo-controlled, observer-blind, safety and dose-finding Phase Ib/IIa study. This study will evaluate up to four dose levels of the BNT164 investigational vaccines (BNT164a1 and BNT164b1) to select a safe and tolerable dose in a three-dose schedule.

This study includes: Part A (Phase Ib) and Part B (Phase IIa).

DETAILED DESCRIPTION:
In Part A, enrollment for BNT164a1 and BNT164b1 will be conducted independently and in parallel. Part A of the study will enroll participants into four dose groups per investigational medicinal product ([IMP] i.e., BNT164a1 or BNT164b1) who will be stratified by interferon gamma release assay (IGRA) status and then randomized 5:1 for BNT164 (BNT164a1 or BNT164b1):placebo. This part of the study will use a staggered dose escalation schema, i.e., enrollment into the next higher dose level is done sequentially and subject to safety data from the previous dose levels, with sentinel participants for Dose 1 in all dose groups.

Part B of this study is a safety expansion in human immunodeficiency virus (HIV)-negative participants of up to two dose groups per IMP (BNT164a1 or BNT164b1) + placebo selected based on the safety and immunogenicity data from Part A. Participants will be randomized 3:3:3:3:1 to up to four dose groups of BNT164 (BNT164a1 or BNT164b1):placebo.

In both Part A and Part B, participants will undergo a three-dose injection schedule with approximately 8 weeks between the first and second dose and approximately 16 weeks between the second and third dose.

ELIGIBILITY:
Inclusion Criteria (applicable to Part A and Part B unless otherwise specified):

* Have given informed consent by signing and dating an informed consent form before initiation of any study-specific procedures.
* Are 18 to 55 years of age inclusive (in Part A) or 18 years of age or older (in Part B) and have a body mass index over 18.5 kg/m^2 and under 35 kg/m^2 and weigh at least 50 kg.
* Are willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions, and other requirements of the study. This includes that they are able to understand and follow study-related instructions.
* In Part A only: Have a reported history or evidence of (scar) of Bacillus Calmette-Guérin (BCG) vaccination.
* Are overall healthy in the clinical judgment of the investigator based on the medical history and clinical assessment (including physical examination, vital signs, clinical laboratory tests, and 12-lead electrocardiogram [ECG]).
* Hemoglobin ≥12.0 g/dL (in Part A) and ≥11.0 g/dL (in Part B) for volunteers who were born female, ≥13.0 g/dL (in Part A) and ≥12.5 g/dL (in Part B) for volunteers who were born male.
* Volunteers of childbearing potential (VOCBP) must have a negative serum beta-human chorionic gonadotropin pregnancy test at Visit 0 and negative urine pregnancy test results before each IMP administration. Volunteers born female that are postmenopausal (confirmed by follicle stimulating hormone) or permanently sterilized (verified by medical records) will not be considered VOCBP.
* VOCBP who agree to practice a highly effective form of contraception and to require their male partners to use condoms, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this study.
* VOCBP who agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during study, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this study.
* Men who are sexually active with a partner of childbearing potential and have not had a vasectomy who agree to use condoms and to ask their sexual partners to practice a highly effective form of contraception during the study, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this study.
* Men who are willing to refrain from sperm donation, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this study.

Exclusion Criteria (applicable to Part A and Part B unless otherwise specified):

* Any existing condition which may affect vaccine injection and/or assessment of local reactions assessment at the injection site, e.g., tattoos, severe scars, etc.
* Any bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Baseline clinical screening questionnaire positive for pulmonary TB disease or history of sputum sample positive for TB, or history of treatment for TB infection or disease.
* Current febrile illness (body temperature ≥38.0°C) or other acute illness at Visit 0.
* Current or history of the following medical conditions:

  1. Cardiovascular diseases, e.g., myocardial infarction, congestive heart failure, cardiomyopathy, or clinically significant arrhythmias, myocarditis, or pericarditis.
  2. Hypertension

     * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well controlled blood pressure is defined as consistently ≤140 mm Hg systolic and ≤90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤150 mm Hg systolic and ≤90 mm Hg diastolic at enrollment.
     * If a person does not have a history of elevated blood pressure or hypertension previously or during screening, also exclude for systolic blood pressure ≥150 mm Hg at enrollment or diastolic blood pressure ≥100 mm Hg at enrollment.
  3. Diabetes mellitus type 1 or type 2 cases requiring medication.
  4. Thyroidectomy, or thyroid disease requiring medication during the last 12 months.
  5. Malignancy within 5 years of Visit 0, excluding localized basal or squamous cell cancer.
  6. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), or (in Part B only) are on a medication determined by the investigator to increase the risk of bleeding.
  7. Seizure disorder: History of seizure(s) within past 3 years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
  8. An abnormal screening or Visit 1 ECG (i.e., showing the corrected QT interval by Fridericia (QTcF) >450 ms; significant ST-T wave changes suggestive of myocardial ischemia or of an acute or indeterminate-age myocardial infarction; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions; complete right or left bundle branch block [QRS >120 ms]; second- or third-degree atrioventricular block); or other clinically significant abnormalities on the ECG at the investigator's discretion.
* History of syncope (fainting) in association with administration of injectable vaccines.
* Known or suspected immunodeficiency.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study IMP.
* Positive test result at Visit 0 or history of hepatitis B, hepatitis C, or HIV.
* History of previous administration of experimental TB vaccines, or any planned non-study vaccinations within 28 days before Dose 1 and continuously until 28 days after Dose 3 (Visit 11).

  * Note: Licensed vaccines are allowed to be given at least 28 days before or 28 days after each IMP administration.
* Current or planned treatment with immunosuppressive therapy, including systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥5 mg/day of prednisone or equivalent) starting at Visit 0 and continuously until 28 days after Dose 3 (Visit 11), for an autoimmune disease. Intraarticular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Have received/donated or plan to receive/donate blood/plasma products or immunoglobulin from 120 days before Dose 1 and continuously until 28 days after Dose 3 (Visit 11).
* Use of any non-study IMP within 28 days before Dose 1 in this study (Visit 1) or planned receipt continuously until Visit 14 in this study (in Part A) or until the end of study visit in this study (Part B), or participate in the active treatment phase of another interventional clinical study.
* Are subject to exclusion periods from another investigational clinical study.
* Are breastfeeding or are planning pregnancy within 90 days after Dose 3 in this study or to father children during the study or within 90 days after Dose 3 in this study.
* Any screening hematology and/or blood chemistry laboratory value that meets the definition of a Grade ≥1 abnormality (in Part A) and of a Grade >1 abnormality (in Part B) at Visit 0 according to the US Food and Drug Administration toxicity grading guidance. For laboratory values for which toxicity grading guidance is not available, participant eligibility will be determined at the discretion of the investigator.

  * Note: Study participants with any stable Grade 1 abnormalities (in Part A) or Grade ≤1 abnormalities (Part B) (according to the toxicity grading scale) may be considered eligible at the discretion of the investigator. For Part A only: A "stable" Grade 1 laboratory abnormality is defined as a report of Grade 1 on an initial blood sample that remains Grade ≤1 upon repeat testing on a second sample from the same participant.
* History of psychiatric illness, including alcohol abuse or drug addiction within 1 year before Visit 0, or a history (within the past 5 years) of substance abuse or known medical, psychological, or social conditions which, in the opinion of the investigator, could compromise their wellbeing if they participate as participants in the study, or that could prevent, limit, or confound the protocol specified assessments.
* Are vulnerable individuals as per International Council on Harmonisation E6 definition, i.e., are individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. This includes investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
* IGRA status at Visit 0 is negative or positive and enrollment for the respective IGRA-negative or IGRA-positive stratum has already been reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited local reactions (pain, erythema/redness, induration/swelling) at the injection site up to 7 days after each dose | Up to 7 days after each dose
  Part A and Part B
Frequency of solicited systemic reactions (vomiting, diarrhea, headache, fatigue, muscle pain & joint pain, chills, and fever) up to 7 days after each dose | Up to 7 days after each dose
  Part A and Part B
Proportion of participants with at least one adverse event (AE) occurring from each dose to 28 days after each dose | From each dose up to 28 days after each dose
  Part A and Part B
Proportion of participants with at least one unsolicited AE occurring from Dose 1 to 28 days post-Dose 3 | From Dose 1 up to 28 days post-Dose 3
  Part A and Part B
Proportion of participants with at least one serious AE or AE of special interest occurring from Dose 1 up to 168 days post-Dose 3 | From Dose 1 up to 168 days post-Dose 3
  Part A and Part B. In Part A, from Dose 1 up to 168 days post-Dose 3. In Part B, from Dose 1 up to 28 days post- Dose 3.
Number of unsolicited AEs from Dose 1 to 28 days post-Dose 3 | From Dose 1 up to 28 days post-Dose 3
  Part A and Part B

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (8):
- Mozambique (2):
  - Centro de Investigação em Saúde de Manhiça (CISM) (recruiting participants for Part B only), Manhiça
  - Centro de Investigação e Treino em Saúde da Polana Caniço (CISPOC) (recruiting participants for Part B only), Maputo
- South Africa (6):
  - CAPRISA eThekweni Clinical Research Site, Berea
  - South African Tuberculosis Vaccine Initiative SATVI, Cape Town
  - Centre for Lung Infection and Immunity UCT Lung Institute, Cape Town
  - Desmond Tutu Health Foundation - Masiphumele Research Office, Cape Town
  - Africa Health Research Institute (AHRI), Mtubatuba
  - The Aurum Institute Tembisa CRC Clinic 4, Tembisa

IPD SHARING:
Plan to Share IPD: No